CLINICAL TRIAL: NCT00398060
Title: GOAL Life-Style Change Implementation Intervention to Prevent Type 2 Diabetes in Primary Health Care
Brief Title: GOAL Life-Style Change Intervention to Prevent Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Academy of Finland (Other)
Responsible Party: Senior researcher Pilvikki Absetz, National Public Health Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KTL223-3
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2008-02

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: life-style counseling; type 2 diabetes; prediabetes; physical activity; diet; cognitive-behavioral
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Prediabetic State; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: Cognitive-behavioral life-style counseling

INTERVENTIONS:
Behavioral: Cognitive-behavioral life-style counseling

SUMMARY:
Life-style change achieved in controlled experimental condition has been shown to prevent type 2 diabetes. The purpose of this study is to evaluate to what extent the life-style change can be achieved in a routine health care setting.

DETAILED DESCRIPTION:
The GOAL (Good Ageing in Lahti region) Program Life-style change implementation trial to prevent type 2 diabetes was set to examine and enhance the effectiveness of life-style change counselling in the primary health care. In the intervention, specific nutritional, physical activity and weight loss objectives shown effective in diabetes prevention in an earlier randomised controlled trial are used as a benchmark, embedded in a structured group counselling model with an empowerment-oriented approach and adapted into the primary health care setting. In the trial, effectiveness and process are evaluated, the analyses including gender and socio-economic differences. Participants were 361 middle-aged (50-65 yrs) adults at an increased risk for type 2 diabetes, recruited in 16 primary health care centres in Paijat-Hame, Finland. Intervention and data collection took place in year 2003.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes risk test score > 11 (Lindstrom & Tuomilehto, 2003)

Exclusion Criteria:

* mental health problem or substance abuse likely to interfere with participation
* acute cancer
* type 2 diabetes requiring pharmacological treatment
* myocardial infarction during the past six months

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2003-01; Primary Completion 2004-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Nutrition (fat, fiber) | 0-1 years
Physical activity | 0-3 years
Weight | 0-3 years

SECONDARY OUTCOMES:
Waist circumference | 0-3 years
Plasma glucose (fasting, 2 hr challenge) | 0-3 years
Serum lipids | 0-3 years
Blood pressure (diastolic, systolic) | 0-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Antti Uutela, PhD, Study Director — National Public Health Institute; Pilvikki Absetz, PhD, Principal Investigator — National Public Health Institute; Martti Talja, PhD, Study Director — Päijät Häme Central Hospital
Locations (1):
- Päijät-Häme Hospital District, Lahti, Finland

REFERENCES:
- [Background] Uutela A, Absetz P, Nissinen A, Valve R, Talja M, Fogelholm M. Health psychological theory in promoting population health in Paijat-Hame, Finland: first steps toward a type 2 diabetes prevention study. J Health Psychol. 2004 Jan;9(1):73-84. doi: 10.1177/1359105304036103. PMID 14683570